CLINICAL TRIAL: NCT07192978
Title: Does Preoperative Physical Activity Predict Postoperative Complications After Incisional Hernia Repair ?
Acronym: EVENTEST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9768
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Incisional Hernia
Keywords: Incisional Hernia; Laparotomy; Comprehensive Complication Index; Clavien-Dindo classification
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with abdominal wall incisional hernia often have numerous comorbidities, making management complex.

To date, no study has described the relationship between preoperative physical activity and the occurrence of complications, particularly severe ones, after incisional hernia repair.

The research hypothesis is that "patient fragility" related to physical inactivity and comorbidities is a poor prognostic factor for the occurrence of complications after incisional hernia repair and a source of more severe complications.

ELIGIBILITY:
Inclusion Criteria

* Adult (≥18 years old)
* Subject operated on at the HUS between January 6, 2021 and October 24, 2024
* Midline eventration
* Placement of a prosthetic reinforcement

Exclusion Criteria

- Subject (and/or their legal representative, if applicable) who has expressed their opposition to the reuse of their data for scientific research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) operated on at the HUS between January 6, 2021 and October 24, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Complications according to the Comprehensive Complication Index (CCI) | Day 1 postoperatively
  The Comprehensive Complication Index (CCI) Score takes into account all postoperative complications and allows them to be expressed by a score ranging from 0 (no complications) to 100 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de cchirurgie générale & digestive - CHU de Strasbourg - France, Strasbourg, France